CLINICAL TRIAL: NCT06364605
Title: MySpace: the Role of Vision on Perceptual Space Representation
Brief Title: MySpace: the Role of Vision in Representing Space
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIT_UVIP_MySpace
Record Dates: First submitted 2024-03-26; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Blindness; Visual Impairment
Keywords: blindness; infants; spatial representations; EEG; child development; medical device
MeSH Terms: conditions — Blindness; Vision Disorders | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iReach Device Group (Experimental)
  Interventions: Device: Rehabilitation with the iReach novel multisensory medical device

INTERVENTIONS:
Device: Rehabilitation with the iReach novel multisensory medical device — From the results of Phases 1,2 and 3, in Phase 4 a medical device for spatial and sensorimotor rehabilitation in infants aged 3 to 36 months will be tested and developed.

SUMMARY:
My Space aims to identify the ontogenesis of spatial representation through cross-sectional and longitudinal studies in infants, children, and adolescents with typical and atypical development (visual impairments). The results will serve for the design and development of a novel multisensory device for sensorimotor rehabilitation in blind children from the early stages of life.

DETAILED DESCRIPTION:
MySpace is an interventional neuropsychology study purely for scientific purposes, with no diagnostic or therapeutic aims. The project aims to define the role of vision in generating uni- and multi-sensory spatial representations (audio/tactile), essential for proper interaction with the surrounding environment. The project will focus on studying spatial deficits and reorganization mechanisms present in the absence of vision from the early years of development. The results will allow drawing overall conclusions on how we perceive the world and develop rehabilitative protocols to improve the quality of life of individuals with visual sensory disabilities. In detail, the project is divided into 4 macro-objectives:

* Study of the role of vision in the development of uni-sensory spatial representations (Phase 1) through experimental procedures at the behavioral and cortical levels. This phase aims to understand the specific temporal windows within which auditory and tactile spatial representations develop in visually impaired children. This phase involves infants and children in an age range from 3 months to 16 years old, with typical and atypical development (visual disabilities), as well as sighted adults and those with visual disabilities. This phase includes the use of behavioral, kinematic, and neurophysiological techniques, employing EEG systems, to provide an assessment of a participant's response to sensory stimuli. Number of participants: 50 sighted adults, 20 blind adults, 60 blind children, 100 sighted children;
* Role of vision in the development of multi-sensory spatial representations (Phase 2) The objective of Phase 2 is to define, the role of vision in the generation of audio-tactile multi-sensory representations. In this phase, both infants and children ranging from 3 months to 16 years old, with and without visual disabilities, as well as adults with and without visual disabilities, will participate. In Phase 2, experiments will be conducted using behavioral, psychophysical, and motion tracking methods. The neurophysiological architecture associated with multi-sensory integration will be studied using EEG. Number of participants: 80 sighted adults, 20 blind adults, 60 blind children, 120 sighted children;
* Neuro-imaging of spatial representation (Phase 3) Phase 3 will study the mechanisms of cortical reorganization following the absence of vision in the early years of life, particularly those concerning the visual cortex responsible for processing spatial information. This phase involves a single setup in which both adults and children ranging from 3 months to 16 years old take part. This phase hypothesizes that structural changes resulting from a visual disability may emerge during the early years of life when spatial perceptual abilities develop and cortical reorganization begins. In this phase, each participant will undergo structural MRI recording to investigate the structural changes observed during growth in both typical cases and cases of visual disability. Number of participants: 50 sighted adults, 20 blind adults, 30 blind children, 30 sighted children;
* Multi-sensory training (Phase 4) The objective of Phase 4 is the development and evaluation of multi-sensory training aimed at helping visually impaired children improve their spatial representation ability and overcome limitations due to the absence of vision. This phase involves infants with both typical and atypical development (i.e., visual disabilities) aged between 3 and 36 months of life. Experimental sessions will be conducted partly at home and partly in clinical centers participating in the project. Non-invasive and painless auditory and tactile stimuli will be employed, which may come from devices applied to the child's body or from sound-producing objects placed in the environment. For data analysis, video recordings will be carried out, and motion-tracking procedures will be employed. To assess the effectiveness of the training, children will be retested approximately 4 months after the end of the training, following the procedures outlined in Phases 1 and 2. These evaluative sessions will help understand if the effects of rehabilitation persist over time. Additionally, during the initial and final phases of the training, and in the follow-up, EEG techniques will be used to assess any changes in cortical activation due to the training. Number of participants:55 blind children, 55 sighted children.

The preliminary data will utilize the Power Analysis method to calculate the minimum sample size required to achieve a correct effect size for a given dimension. The data will be analyzed using both parametric and non-parametric tests, and differences between groups will be assessed with t-tests, ANOVA, TANCOVA, and linear mixed models where appropriate. An appropriate post-hoc test will be conducted if significance is found. The significance level will be considered at p<0.05. Where necessary, parametric techniques will be replaced by non-parametric equivalents. The standard software used will include: Matlab, R, Origin, Statistica, and SPSS, recognized in the research field. For the analysis of electroencephalographic data, EEGlab and/or Fieldtrip toolboxes will be utilized. For functional magnetic resonance imaging data analysis, the FSL and/or SPM toolboxes will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Having provided (by the subject or the parent/guardian) consent to be contacted through one of the recruitment channels established by the Italian Institute of Technology or voluntary enrollment;
* Signature of the informed consent (by the subject or the parent/guardian);
* Absence of other disabilities/conditions/comorbidities that would prevent participation and/or ensure patient safety during the execution of the tests and/or guarantee the quality/reliability of the data. This point is acquired through Informed Consent, in the section expressly acknowledging the following reasons for ineligibility to participate in the study: tactile hypersensitivity (specifically assessing equipment tolerance), taking neuroactive drugs and substances and having taken them in the last six months, comorbidity with another pathology;
* Being affected, to the best of their knowledge, by pathologies of the central nervous system, and having experienced epileptic episodes, even minor ones, and convulsive crises in general, even in childhood;
* The participating subjects may have typical or atypical development (i.e., group with visual disability). In the case of visual impairment, the disability should be congenital (from birth) or late onset. Furthermore, the following requirements must be met: subjects with visual disabilities must be classified according to current diagnostic rules, with visual problems present from birth or occurring later, with residual vision ranging from 0.5-1.3 LogMAR in the case of low vision or lower than 1.3 LogMAR in the case of blindness;
* Age range required for each phase and configuration: Blind adults (≥ 18 years old):

Phase 1; Phase 2; Phase 3; Typical adults (≥ 18 years old): Phase 1; Phase 2; Phase 3; Blind minors (3 months < age < 18 years old): All phases; Typical minors (3 months < age < 18 years old): All phases; Adequate cognitive capacity for age. In particular, recognized scales such as the WISC9 scale will be used as a reference parameter to assess cognitive capacity.

Exclusion Criteria:

* Additional disabilities besides visual impairment (e.g., individuals who are both visually and hearing impaired);
* Absence of the signature on the informed consent form or incomplete consent regarding acknowledgment of the incompatibilities for participation in the study;
* IQ values below the threshold of normality according to one of the recognized international scales;
* Preterm birth.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceptual responses to multisensory stimuli | Through study completion, an average of 5 years
  Evaluation of the number of correct responses and reaction times (in seconds), to uni- and multisensory (audio-tactile) stimuli.
Stimuli velocity perception | Through study completion, an average of 5 years
  Estimation of the speed of a moving stimulus (m/s)
Distance stimuli perception | Through study completion, an average of 5 years
  Estimation of the the distance traveled by a moving stimulus (m), along with an estimate of the error made in identifying the endpoint of the stimulus by the participant (m).
Eye movements | Years 3-5
  Eye movements are evaluated in terms of fixation duration (s) and time to first fixation (TTFF) (ms).
Saccade Analysis | Years 3-5
  Estimation of saccade length (pixels)
ERP evaluation and analysis | Through study completion, an average of 5 years
  Evaluation of the Event-Related-Potentials (ERPs) in terms of the number of spikes and their Amplitude (μV);
Power of the cortical activity | Through study completion, an average of 5 years
  Evaluation of power expressed by the alpha band (8-12 Hz) of the EEG recorded in the occipital area (dB).

CONTACTS AND LOCATIONS:
Locations (1):
- Unit For Visually Impaired People, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gori M. Multisensory Integration and Calibration in Children and Adults with and without Sensory and Motor Disabilities. Multisens Res. 2015;28(1-2):71-99. doi: 10.1163/22134808-00002478. PMID 26152053
- [Result] Gori M, Sandini G, Burr D. Development of visuo-auditory integration in space and time. Front Integr Neurosci. 2012 Sep 17;6:77. doi: 10.3389/fnint.2012.00077. eCollection 2012. PMID 23060759
- [Result] Gori M, Sandini G, Martinoli C, Burr DC. Impairment of auditory spatial localization in congenitally blind human subjects. Brain. 2014 Jan;137(Pt 1):288-93. doi: 10.1093/brain/awt311. Epub 2013 Nov 21. PMID 24271326
- [Result] Finocchietti S, Cappagli G, Gori M. Encoding audio motion: spatial impairment in early blind individuals. Front Psychol. 2015 Sep 7;6:1357. doi: 10.3389/fpsyg.2015.01357. eCollection 2015. PMID 26441733
- [Result] Cappagli G, Gori M. Auditory spatial localization: Developmental delay in children with visual impairments. Res Dev Disabil. 2016 Jun-Jul;53-54:391-8. doi: 10.1016/j.ridd.2016.02.019. Epub 2016 Mar 19. PMID 27002960
- [Result] Barutchu A, Crewther DP, Crewther SG. The race that precedes coactivation: development of multisensory facilitation in children. Dev Sci. 2009 Apr;12(3):464-73. doi: 10.1111/j.1467-7687.2008.00782.x. PMID 19371371
- [Result] Inuggi A, Pichiecchio A, Ciacchini B, Signorini S, Morelli F, Gori M. Multisystemic Increment of Cortical Thickness in Congenital Blind Children. Cereb Cortex Commun. 2020 Oct 9;1(1):tgaa071. doi: 10.1093/texcom/tgaa071. eCollection 2020. PMID 34296131
- [Result] Mongodi S, Ottonello G, Viggiano R, Borrelli P, Orcesi S, Pichiecchio A, Balottin U, Mojoli F, Iotti GA. Ten-year experience with standardized non-operating room anesthesia with Sevoflurane for MRI in children affected by neuropsychiatric disorders. BMC Anesthesiol. 2019 Dec 18;19(1):235. doi: 10.1186/s12871-019-0897-1. PMID 31852450
- [Result] Erden G, Yigit I, Celik C, Guzey M. The diagnostic utility of the Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV) in identification of gifted children. J Gen Psychol. 2022 Jul-Sep;149(3):371-390. doi: 10.1080/00221309.2020.1862038. Epub 2020 Dec 22. PMID 33350363
- [Result] Lawrence A, Choe DE. Mobile Media and Young Children's Cognitive Skills: A Review. Acad Pediatr. 2021 Aug;21(6):996-1000. doi: 10.1016/j.acap.2021.01.007. Epub 2021 Jan 21. PMID 33486100
- [Result] Cappagli G, Cocchi E, Gori M. Auditory and proprioceptive spatial impairments in blind children and adults. Dev Sci. 2017 May;20(3). doi: 10.1111/desc.12374. Epub 2015 Nov 27. PMID 26613827
- [Result] Vercillo T, Burr D, Sandini G, Gori M. Children do not recalibrate motor-sensory temporal order after exposure to delayed sensory feedback. Dev Sci. 2015 Sep;18(5):703-12. doi: 10.1111/desc.12247. Epub 2014 Nov 28. PMID 25444457
- [Result] Tonelli A, Brayda L, Gori M. Task-dependent calibration of auditory spatial perception through environmental visual observation. Front Syst Neurosci. 2015 Jun 2;9:84. doi: 10.3389/fnsys.2015.00084. eCollection 2015. PMID 26082692
- [Result] Cuturi LF, Gori M. The Effect of Visual Experience on Perceived Haptic Verticality When Tilted in the Roll Plane. Front Neurosci. 2017 Dec 6;11:687. doi: 10.3389/fnins.2017.00687. eCollection 2017. PMID 29270109
- [Result] Aggius-Vella E, Campus C, Finocchietti S, Gori M. Audio Spatial Representation Around the Body. Front Psychol. 2017 Nov 3;8:1932. doi: 10.3389/fpsyg.2017.01932. eCollection 2017. PMID 29249999
- [Result] Campus C, Sandini G, Concetta Morrone M, Gori M. Spatial localization of sound elicits early responses from occipital visual cortex in humans. Sci Rep. 2017 Sep 5;7(1):10415. doi: 10.1038/s41598-017-09142-z. PMID 28874681
- [Result] Campus C, Brayda L, De Carli F, Chellali R, Fama F, Bruzzo C, Lucagrossi L, Rodriguez G. Tactile exploration of virtual objects for blind and sighted people: the role of beta 1 EEG band in sensory substitution and supramodal mental mapping. J Neurophysiol. 2012 May;107(10):2713-29. doi: 10.1152/jn.00624.2011. Epub 2012 Feb 15. PMID 22338024
- [Result] Rigato S, Begum Ali J, van Velzen J, Bremner AJ. The neural basis of somatosensory remapping develops in human infancy. Curr Biol. 2014 Jun 2;24(11):1222-6. doi: 10.1016/j.cub.2014.04.004. Epub 2014 May 22. PMID 24856214
- [Result] Klostermann A, Hossner EJ. The Quiet Eye and Motor Expertise: Explaining the "Efficiency Paradox". Front Psychol. 2018 Feb 8;9:104. doi: 10.3389/fpsyg.2018.00104. eCollection 2018. PMID 29472882
- [Result] Richmond J, Nelson CA. Relational memory during infancy: evidence from eye tracking. Dev Sci. 2009 Jul;12(4):549-56. doi: 10.1111/j.1467-7687.2009.00795.x. PMID 19635082
- [Result] Stoll J, Chatelle C, Carter O, Koch C, Laureys S, Einhauser W. Pupil responses allow communication in locked-in syndrome patients. Curr Biol. 2013 Aug 5;23(15):R647-8. doi: 10.1016/j.cub.2013.06.011. PMID 23928079
- [Result] Takacs ZK, Bus AG. Benefits of Motion in Animated Storybooks for Children's Visual Attention and Story Comprehension. An Eye-Tracking Study. Front Psychol. 2016 Oct 13;7:1591. doi: 10.3389/fpsyg.2016.01591. eCollection 2016. PMID 27790183
- [Result] Delorme A, Makeig S. EEGLAB: an open source toolbox for analysis of single-trial EEG dynamics including independent component analysis. J Neurosci Methods. 2004 Mar 15;134(1):9-21. doi: 10.1016/j.jneumeth.2003.10.009. PMID 15102499